CLINICAL TRIAL: NCT01021553
Title: A Phase II Study to Evaluate: Delay in Intravaginal Ejaculatory Latency Time (IELT), Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Two Oral Doses of GSK557296 in a Randomized, Double Blind, Placebo-Controlled, Parallel Group Study in Men With Premature Ejaculation
Brief Title: A Study To Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Two Oral Doses of GSK557296 in a Study in Men With Premature Ejaculation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109059
Record Dates: First submitted 2009-11-12; First posted 2009-11-30 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Premature Ejaculation
Keywords: Proof of Concept; Double Blind
MeSH Terms: conditions — Premature Ejaculation | interventions — epelsiban; MG 50-3-1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- 50 mg (Active Comparator): 50 mg GSK557296
  Interventions: Drug: GSK557296
- 150 mg (Active Comparator): 150 mg GSK557296
  Interventions: Drug: GSK557296

INTERVENTIONS:
Drug: GSK557296 — 50 mg GSK557296
  Other Names: 50 mg
  Arms: 50 mg
Drug: GSK557296 — 150 mg GSK557296
  Other Names: 150 mg
  Arms: 150 mg
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
To determine if an on demand dosing of 50 mg or 150 mg of GSK557296 demonstrates superior efficacy with respect to duration of intra vaginal ejaculatory latency time (IELT) during an 8 week study period compared to placebo in men with primary premature ejaculation. An assessment of the safety and tolerability of all doses of GSK557296 will be performed as well as an assessment for change in the Index of Premature Ejaculation (IPE) from baseline and at the end of the 8 weeks of treatment. During the active treatment period study participants will be limited to a maximum of 40 doses of GSK557296, or placebo, spilt as 20 doses for both 4 week intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Males with primary PE, according to the ISSM Consensus Definition. Defined as, a male sexual dysfunction characterized by ejaculation which always or nearly always occurs prior to or within about one minute of vaginal penetration; and, inability to delay ejaculation on all or nearly all vaginal penetrations; and, negative personal consequences, such as distress, bother, frustration and/or the avoidance of sexual intimacy
2. Stable heterosexual relationship, with a single non pregnant, nonlactating female partner using adequate contraception (as confirmed by oral questioning of male study subject) in a relationship of greater than >4 months duration. This same partner will be the one with whom the subject makes and records all IELT attempts during the duration of the study.
3. Aged between 18 and 50 years (i.e. subjects must not have completed their 50th year birthday at the time of screening, but can turn 50 years during the course of the study).
4. The subject must make at least four attempts at sexual intercourse on four separate days during the untreated run in period.
5. The average intravaginal ejaculatory latency time must be <65 seconds based on the study-provided stop watch assessments

Exclusion Criteria:

1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result and positive HIV antibody and or confirmatory ELISA test at screening.
2. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).

Previous or Current Medical Conditions

1. Erectile dysfunction (defined as IIEF-EF domain score < 22)
2. Active or recent (< 6 months) history of prostatitis, as determined by patient symptoms or treatment seeking for newly diagnosed or flare of symptoms related to previously diagnosed prostatitis.
3. Any unstable medical, psychiatric or substance abuse disorder that in the opinion of the investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study.
4. Presence of penile anatomical abnormalities (e.g. penile fibrosis or Peyronie's disease) that in the opinion of the investigator would significantly impair sexual performance.
5. Prior implantation of penile implant for erectile dysfunction
6. Primary hypoactive sexual desire.
7. Spinal cord injury.
8. History of seizures, within last 6 months.
9. History of prostate cancer treated or untreated.
10. History of prostatectomy or prostate procedures for any cause.
11. Clinically significant chronic hematological disease which may lead to priapism such as sickle cell anemia, multiple myeloma or leukemia.
12. Significant active peptic ulceration.
13. Presence of the following conditions prior to screening: myocardial infarction, coronary bypass surgery, coronary artery angioplasty, unstable angina, clinically evident congestive heart failure, cardiac pacemaker, or cerebrovascular accident.
14. Cardiac arrhythmia: significant cardiac arrhythmia shown on screening ECG, or a known or suspected history of significant cardiac arrhythmias within six months prior to screening. i.e., pre-existing syndromes, sinus pause > 3 seconds, non-sustained ventricular tachycardia (3 consecutive ectopic beats), sustained ventricular tachycardia (30 consecutive ectopic beats), sustained supraventricular tachycardia (30 consecutive ectopic beats), accessory pathway tachycardia, bradycardia (heart rate < 50 beats per minute), atrial flutter, atrial fibrillation, ectopic pacemaker, sick sinus syndrome, ventricular block (second or third degree), or bundle branch block. Uncontrolled atrial fibrillation/flutter (ventricular response rate less than or equal to 100 bpm) at the screening visit (Visit 1).
15. History of congenital QT prolongation and/or QTc interval >450msec at screening visit (Visit 1) using the Bazett formula.
16. Mean systolic cuff BP > 140 mmHg, as assessed by three measurements taken in sequence within 5-10ming of last measure. Taken with the study subject in a supine position at the screening visit (Visit 1).
17. Mean diastolic cuff BP >90 mmHg, as assess by three measurements taken in sequence within 5-10 minutes of the last measure. Taken with the study subject in a supine position at the screening visit (Visit 1).
18. History of malignancy within the past five years (other than squamous or basal cell skin cancer).
19. Any condition which would preclude sexual activity.

Concomitant Medications

1. No concomitant medications maybe used within 7 days of Visit 1 and or at any time during the study including oral medications, vacuum devices, constrictive devices, injections, urethral suppositories, gels, any over-the-counter herbal or non-prescription medications, and products purchased via the internet or mail order pharmacies. During the course of the study concomitant medication use can be considered upon consultation and prior agreement with primary investigator and medical monitor. Specific exceptions for asthmatic patients and patients with allergic rhinitis, who are on stable doses of inhaled or intra nasal agents as prescribed by their health care providers, and who have had no adjustments in their prescribed and or actual use within the last 60 days. Agents which are known or expected to have significant systemic exposures as a result of inhaled or intra-nasal use or to have known CYP3A4 drug-drug interaction potential are not included in this exemption.
2. Subjects who have received any investigational drug (including placebo) within 30 days of the screening visit or 5 half lives of the investigational drug whichever is longer (Visit 1).

Abnormal Laboratory Values

1. Subjects who have a serum total testosterone level >25% below the lower limit of normal according to the range of the testing laboratory, when obtained in the morning versus in the afternoon, from screening lab which will need to be evaluated prior to randomization.
2. Subjects with a clinically significant elevation of serum creatinine of > 2.0 when obtained from a screening lab which will need to be evaluated prior to randomization.
3. Subject with a clinically significant elevation of AST of > 126 and/or ALT of > 144 when obtained from a screening lab which will need to be evaluated prior to randomization.
4. Screening PSA > 4.0 ng/ml
5. TSH outside the normal reference ranges at visit 1
6. Free Triiodothyronine [T3] outside the normal reference ranges at visit 1
7. Free Thyroxine T4 outside the normal reference ranges at visit 1

Other exclusion criteria

1. Severe chronic or acute liver disease, history of moderate (Child-Pugh B) or severe (Child-Pugh C) hepatic impairment.
2. Subjects with known hypersensitivity to GSK557296 or any component of the investigational medication.
3. Subjects who are illiterate or unable to understand the questionnaires or the subject diary.
4. Subjects who are unwilling or unable to complete the subject diary.
5. Subjects who are unwilling to be randomized to placebo.
6. Subject whose sexual partner is actively trying to conceive, and or is unwilling to use a reliable form of birth control as outlined in Section 8.1 for the duration of the trial. Or whose female partner is breast feeding.
7. Subjects, who in the opinion of the investigator, would be non-compliant with the majority of the visits scheduled or study procedures.
8. History of sensitivity to heparin or heparin-induced thrombocytopenia (for subjects at sites where PK studies are planned).
9. Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 1 month prior to screening.
10. Consumption of seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication, and for the duration of the study.
11. Subjects who have consumed alcohol within 24 hours will have their PK session rescheduled.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2009-12-23 (Actual); Primary Completion 2011-05-05 (Actual); Study Completion 2011-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (6):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Bala-Cynwyd, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Shinghal R, Barnes A, Mahar KM, Stier B, Giancaterino L, Condreay LD, Black L, McCallum SW. Safety and efficacy of epelsiban in the treatment of men with premature ejaculation: a randomized, double-blind, placebo-controlled, fixed-dose study. J Sex Med. 2013 Oct;10(10):2506-17. doi: 10.1111/jsm.12272. Epub 2013 Aug 12. PMID 23937679
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 109059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109059 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 sites in United States and 2 centers in the Netherlands during 23 December 2009 to 05 May 2011.
Pre-assignment Details: The study consisted of 4 weeks run-in period. Total 77 male participants with primary pre-mature ejaculation were enrolled and randomized. Out of these 65 participants completed the study.
Groups:
- Placebo: Participants received 3 placebo tablets matching study drug approximately one hour prior to planned sexual intercourse (SI), once in a 24-hour time period, on-demand for 8 weeks.
- GSK557296 50 mg: Participants received one 50 milligrams (mg) tablet of study drug and two placebo tablets approximately one hour prior to planned SI, once in a 24-hour time period, on-demand for 8 weeks.
- GSK557296 150 mg: Participants received three 50 mg tablets of study drug approximately one hour prior to planned SI, once in a 24-hour time period, on-demand for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg
Started | 27 | 22 | 28
Completed | 23 | 17 | 25
Not Completed | 4 | 5 | 3
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 2 | 0
Not completed — Protocol Violation | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received 3 tablets approximately one hour prior to planned SI, once in a 24-hour time period, on-demand for 8 weeks.
- GSK557296 50 mg: Participants received one 50 mg tablet of study drug and two placebo tablets approximately one hour prior to planned SI, once in a 24-hour time period, on-demand for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg | Total
Number analyzed (Participants) | 27 | 22 | 28 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.4 (8.90) | 37.9 (9.85) | 34.0 (9.00) | 36.7 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 27 | 22 | 28 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 2 | 2 | 3 | 7
  White | 24 | 20 | 21 | 65
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Intravaginal Ejaculatory Latency Time (IELT) Compared Over All 8 Weeks of Treatment or Until Premature Discontinuation
Description: Male participant needed to make a minimum of 4 attempts at SI and Baseline IELTs were assessed by stop watch measurements for each SI attempt. IELT was the elapsed time from vaginal penetration until ejaculation. On-treatment IELT for each participant was calculated by taking the median IELT from all valid on-treatment IELT attempts. Geometric mean IELT for each treatment was compared using analysis of covariance (ANCOVA). LS mean values and two-sided p-values are from the general linear model ln(median IELT)= ln(Baseline IELT) + treatment + cluster. A step-down procedure was used to determine if the efficacy of on-demand GSK557296 was superior to placebo. First, the average of the geometric mean IELTs of the pooled 150mg and 50mg doses of GSK557296 was tested against placebo, and if significance was achieved with this global plateau trend test (p < 0.05), then the simultaneous pair wise comparisons of the 150mg and 50mg doses to placebo would occur (each at an alpha level of 0.05).
Time Frame: Up to Week 8
Population: Intent to Treat (ITT) Population consisted of all participants randomized to study treatment. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: minutes
Groups:
- Pooled GSK557296: These were pooled participants population from the groups who received GSK55729650 mg and 150 mg.
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg | Pooled GSK557296
Number analyzed (Participants) | 25 | 20 | 26 | 46
minutes | 0.62 (0.090) | 0.72 (0.117) | 0.69 (0.099) | 0.71 (0.075)
Statistical Analysis 1: Comparison: Placebo vs GSK557296 50 mg; Test type: Superiority or Other; p = 0.4959, ANCOVA; Geometric LS Mean Fold Difference = 1.16, 95% CI 2-sided [0.75 to 1.79] — Estimated value is Geometric LS Mean Fold Difference from Placebo
Statistical Analysis 2: Comparison: Placebo vs GSK557296 150 mg; Test type: Superiority or Other; p = 0.6161, ANCOVA; Geometric LS Mean Fold Difference = 1.11, 95% CI 2-sided [0.74 to 1.65] — Estimated value is Geometric LS Mean Fold Difference from Placebo
Statistical Analysis 3: Comparison: Placebo vs Pooled GSK557296; Test type: Superiority or Other; p = 0.4971, ANCOVA; Geometric LS Mean Fold Difference = 1.13, 95% CI 2-sided [0.79 to 1.61] — Estimated value is Geometric LS Mean Fold Difference from Placebo

2. Secondary Outcome: Mean IELT Compared After Each 4-week Treatment Period, or Until Premature Discontinuation
Description: as for outcome 1
Time Frame: Up to Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: minutes
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg | Pooled GSK557296
Number analyzed (Participants) | 27 | 22 | 28 | 50
minutes
  Week 0 to 4: number analyzed (Participants) | 25 | 20 | 26 | 46
  Week 0 to 4 | 0.67 (0.095) | 0.69 (0.109) | 0.67 (0.094) | 0.68 (0.071)
  Week 4 to 8: number analyzed (Participants) | 23 | 17 | 24 | 41
  Week 4 to 8 | 0.65 (0.110) | 0.86 (0.168) | 0.70 (0.118) | 0.77 (0.097)
Statistical Analysis 1: Comparison: Placebo vs GSK557296 50 mg; For Week 0 to 4; Test type: Superiority or Other; p = 0.9037, ANCOVA; Geometric LS Mean Fold Difference = 1.03, 95% CI 2-sided [0.67 to 1.58] — Estimated value is Geometric LS Mean Fold Difference from Placebo
Statistical Analysis 2: Comparison: Placebo vs GSK557296 150 mg; For Week 0 to 4; Test type: Superiority or Other; p = 0.9939, ANCOVA; Geometric LS Mean Fold Difference = 1.00, 95% CI 2-sided [0.67 to 1.48] — Estimated value is Geometric LS Mean Fold Difference from Placebo
Statistical Analysis 3: Comparison: Placebo vs Pooled GSK557296; For Weeks 0-4; Test type: Superiority or Other; p = 0.9541, ANCOVA; Geometric LS Mean Fold Difference = 1.01, 95% CI 2-sided [0.71 to 1.43] — Estimated value is Geometric LS Mean Fold Difference from Placebo
Statistical Analysis 4: Comparison: Placebo vs GSK557296 50 mg; For Weeks 4-8; Test type: Superiority or Other; p = 0.2798, ANCOVA; Geometric LS Mean Fold Difference = 1.33, 95% CI 2-sided [0.79 to 2.24] — Estimated value is Geometric LS Mean Fold Difference from Placebo
Statistical Analysis 5: Comparison: Placebo vs GSK557296 150 mg; For Weeks 4-8; Test type: Superiority or Other; p = 0.7255, ANCOVA; Geometric LS Mean Fold Difference = 1.09, 95% CI 2-sided [0.68 to 1.75] — Estimated value is Geometric LS Mean Fold Difference from Placebo
Statistical Analysis 6: Comparison: Placebo vs Pooled GSK557296; For Weeks 4-8; Test type: Superiority or Other; p = 0.4347, ANCOVA; Geometric LS Mean Fold Difference = 1.18, 95% CI 2-sided [0.77 to 1.80] — Estimated value is Geometric LS Mean Fold Difference from Placebo

3. Secondary Outcome: Mean IELT Compared After the First Dose of Study Drug or Placebo
Description: Male participants needed to make a minimum of 4 attempts at SI and Baseline IELTs were assessed by stop watch measurements for each SI attempt. IELT was the elapsed time from vaginal penetration until ejaculation. First dose IELT was the IELT value associated with the first valid SI attempt made during the treatment period. For GSK557296 50 mg and 150 mg: LS mean values and two-sided p-values are from the general linear model ln(median IELT)= ln(Baseline IELT) + treatment + cluster using placebo, GSK557296 50 mg and GSK557296 150 mg treatments. A step-down procedure was used to determine if the efficacy of on-demand GSK557296 was superior to placebo. First, the average of the geometric mean IELTs of the pooled 150mg and 50mg doses of GSK557296 was tested against placebo, and if significance was achieved with this global plateau trend test (p < 0.05), then the simultaneous pair wise comparisons of the 150mg and 50mg doses to placebo would occur (each at an alpha level of 0.05).
Time Frame: Up to Week 8
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: minutes
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg | Pooled GSK557296
Number analyzed (Participants) | 25 | 20 | 26 | 46
minutes | 0.60 (0.116) | 0.68 (0.146) | 0.57 (0.109) | 0.61 (0.088)
Statistical Analysis 1: Comparison: Placebo vs GSK557296 50 mg; Test type: Superiority or Other; p = 0.6583, ANCOVA; Geometric LS Mean Fold Difference = 1.14, 95% CI 2-sided [0.63 to 2.05] — Estimated value is Geometric LS Mean Fold Difference from Placebo
Statistical Analysis 2: Comparison: Placebo vs GSK557296 150 mg; Test type: Superiority or Other; p = 0.8790, ANCOVA; Geometric LS Mean Fold Difference = 0.96, 95% CI 2-sided [0.56 to 1.65] — Estimated value is Geometric LS Mean Fold Difference from Placebo
Statistical Analysis 3: Comparison: Placebo vs Pooled GSK557296; Test type: Superiority or Other; p = 0.8971, ANCOVA; Geometric LS Mean Fold Difference = 1.03, 95% CI 2-sided [0.64 to 1.67] — Estimated value is Geometric LS Mean Fold Difference from Placebo

4. Secondary Outcome: Mean Change From Baseline in IELT Compared After Each 4-week Treatment Period and Over All 8 Weeks or Until Premature Discontinuation
Description: Male participants needed to make a minimum of 4 attempts at SI and Baseline IELTs were assessed by stop watch measurements for each SI attempt. IELT was the elapsed time from vaginal penetration until ejaculation. Baseline IELT was calculated as the arithmetic mean IELT from valid screening SI attempts. If multiple screening SI attempts were made on the same calendar day, only the IELT from the first attempt was used in the calculation of Baseline IELT. Change from Baseline IELT was calculated by subtracting the Baseline IELT (arithmetic mean IELT from valid screening attempts) from the on-treatment IELT (median IELT from valid on-treatment attempts). Only participants with a Baseline and a post-Baseline IELT value were included.
Time Frame: Baseline and up to Week 8
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg | Pooled GSK557296
Number analyzed (Participants) | 27 | 22 | 28 | 50
minutes
  Week 0 to 4: number analyzed (Participants) | 25 | 20 | 26 | 46
  Week 0 to 4 | 0.29 (0.510) | 0.74 (2.061) | 1.26 (3.493) | 1.03 (2.939)
  Week 4 to 8: number analyzed (Participants) | 23 | 17 | 24 | 41
  Week 4 to 8 | 0.38 (0.940) | 1.24 (2.869) | 1.30 (2.853) | 1.27 (2.823)
  Week 0 to 8: number analyzed (Participants) | 25 | 20 | 26 | 46
  Week 0 to 8 | 0.26 (0.481) | 0.91 (2.406) | 1.24 (3.085) | 1.10 (2.786)

5. Secondary Outcome: Mean Change From Baseline in IELT Compared After the First Dose of Study Drug or Placebo
Description: Male participants needed to make a minimum of 4 attempts at SI and Baseline IELTs were assessed by stop watch measurements for each SI attempt. IELT was the elapsed time from vaginal penetration until ejaculation. First dose IELT was the IELT value associated with the first valid SI attempt made during the treatment period. Baseline IELT was calculated as the arithmetic mean IELT from valid screening SI attempts. If multiple screening SI attempts were made on the same calendar day, only the IELT from the first attempt was used in the calculation of Baseline IELT. Change from Baseline IELT was calculated by subtracting the Baseline IELT (arithmetic mean IELT from valid screening attempts) from the on-treatment IELT (median IELT from valid on-treatment attempts). Only participant with a Baseline IELT and a valid first attempt were included.
Time Frame: Baseline and Week 4
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg | Pooled GSK557296
Number analyzed (Participants) | 25 | 20 | 26 | 46
minutes | 0.33 (0.750) | 0.73 (2.003) | 0.93 (3.191) | 0.84 (2.713)

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time [AUC(0-inf)] and From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration [AUC(0-t)] of GSK557296
Description: The pharmacokinetic (PK ) visit was not needed to take place at visit 2 but supposed to be completed before visit 3. The participants were asked to fast overnight prior to their PK sampling day and the time of their last meal was recorded.
Time Frame: At 0, 0.25, 0.5, 0.75, 1, 2, 4, 6 and 8 hours at visit 2 or within 7 days of randomization
Population: PK Population consisted of all participants from whom a PK sample had been obtained and analyzed. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours times nanograms per milliliters
Arm/Group | GSK557296 50 mg | GSK557296 150 mg
Number analyzed (Participants) | 21 | 28
Hours times nanograms per milliliters
  AUC (0-inf) | 854.1 (45) | 2485.9 (33)
  AUC (0-t) | 772.9 (43) | 2304.2 (31)
Statistical Analysis 1: Comparison: GSK557296 50 mg vs GSK557296 150 mg; Test type: Superiority or Other; Ratio of treatments = 2.91, 90% CI 2-sided [2.43 to 3.48] — For AUC (0-inf)
Statistical Analysis 2: Comparison: GSK557296 50 mg vs GSK557296 150 mg; Test type: Superiority or Other; Ratio of treatments = 2.98, 90% CI 2-sided [2.51 to 3.54]

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK557296
Description: The PK visit was not needed to take place at visit 2 but supposed to be completed before visit 3. The participants were asked to fast overnight prior to their PK sampling day and the time of their last meal was recorded.
Time Frame: At 0, 0.25, 0.5, 0.75, 1, 2, 4, 6 and 8 hours at visit 2 or within 7 days of randomization
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | GSK557296 50 mg | GSK557296 150 mg
Number analyzed (Participants) | 21 | 28
Nanograms per milliliter (ng/mL) | 387.2 (49) | 1405.1 (41)
Statistical Analysis 1: Comparison: GSK557296 50 mg vs GSK557296 150 mg; Test type: Superiority or Other; Ratio of treatments = 3.63, 90% CI 2-sided [2.95 to 4.47]

8. Secondary Outcome: Time of Occurrence of Maximum Observed Plasma Concentration (Tmax) of GSK557296
Description: as for outcome 7
Time Frame: At 0, 0.25, 0.5, 0.75, 1, 2, 4, 6 and 8 hours at visit 2 or within 7 days of randomization
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | GSK557296 50 mg | GSK557296 150 mg
Number analyzed (Participants) | 21 | 28
hours | 0.6 (43) | 0.4 (51)

9. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were taken in a seated position. If the single measure was outside the cut off value, the mean of three seated measures were taken approximately 5-10 minutes apart was recorded. Baseline value was the latest values obtained on or before the Baseline reference date. Change from Baseline was the value at any visit post-Baseline minus value at Baseline. Per-participant values for all vital sign measures were taken as the mean of all reported values on a given date, regardless of recorded position.
Time Frame: Baseline and up to follow up (post treatment 48 hours)
Population: The Safety Population consisted of all participants randomized to study treatment who received at least one dose of study drug. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg
Number analyzed (Participants) | 25 | 22 | 28
Millimeters of mercury
  SBP, Week 4: number analyzed (Participants) | 25 | 21 | 27
  SBP, Week 4 | 0.422 (8.5478) | -2.472 (9.3388) | -0.550 (8.8500)
  SBP, Week 8: number analyzed (Participants) | 23 | 17 | 25
  SBP, Week 8 | 1.290 (9.1774) | -0.657 (11.1552) | -4.268 (13.4694)
  DBP, Week 4: number analyzed (Participants) | 25 | 21 | 27
  DBP, Week 4 | -0.226 (7.5436) | -2.036 (7.3751) | -0.485 (6.7274)
  DBP, Week 8: number analyzed (Participants) | 23 | 17 | 25
  DBP, Week 8 | 0.188 (7.8127) | 1.529 (6.9245) | -0.897 (8.8300)

10. Secondary Outcome: Mean Change From Baseline in Heart Rate
Description: Heart rate assessment was done in a seated position. If the single measure was outside the cut off value, the mean of three seated measures were taken approximately 5-10 minutes apart was recorded. Baseline value was the latest values obtained on or before the Baseline reference date. Change from Baseline was the value at any visit post-Baseline minus value at Baseline. Per-participant values for all vital sign measures were taken as the mean of all reported values on a given date, regardless of recorded position.
Time Frame: Baseline and up to follow up (post treatment 48 hours)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg
Number analyzed (Participants) | 25 | 22 | 28
Beats per minute
  Week 4: number analyzed (Participants) | 25 | 21 | 27
  Week 4 | 0.319 (8.4404) | 1.821 (10.5332) | 3.240 (9.8555)
  Week 8: number analyzed (Participants) | 23 | 17 | 25
  Week 8 | 2.428 (6.9642) | 2.221 (6.2480) | 0.279 (7.8860)

11. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Values
Description: ECG parameter values for QT interval, QT duration corrected for heart rate by Fridericia's formula (QTc [Fridericia]), QT duration corrected for heart rate by Bazett's formula (QTc [Bazett]), PR Interval and QRS Duration were assessed. The Baseline ECG was the latest ECG recorded on or before the participant's Baseline reference date. Change from Baseline was the value at any visit post-Baseline minus value at Baseline.
Time Frame: Baseline and up to follow up (post treatment 48 hours)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg
Number analyzed (Participants) | 25 | 22 | 28
Milliseconds
  QT Interval, Week 4: number analyzed (Participants) | 25 | 21 | 27
  QT Interval, Week 4 | 1.8 (19.52) | -2.5 (25.42) | -0.1 (21.35)
  QT Interval, Week 8: number analyzed (Participants) | 23 | 17 | 25
  QT Interval, Week 8 | -3.1 (17.16) | -0.4 (20.17) | -4.9 (21.12)
  QTc (Fridericia), Week 4: number analyzed (Participants) | 10 | 7 | 10
  QTc (Fridericia), Week 4 | 1.5 (11.98) | -3.1 (12.77) | -9.2 (13.18)
  QTc (Fridericia), Week 8: number analyzed (Participants) | 10 | 5 | 10
  QTc (Fridericia), Week 8 | -5.7 (8.07) | 5.4 (7.23) | -3.6 (17.42)
  QTc (Bazett), Week 4: number analyzed (Participants) | 25 | 21 | 26
  QTc (Bazett), Week 4 | 0.4 (18.50) | -1.0 (15.80) | -4.2 (16.07)
  QTc (Bazett), Week 8: number analyzed (Participants) | 23 | 17 | 25
  QTc (Bazett), Week 8 | -1.7 (15.88) | 3.4 (17.52) | -4.2 (17.38)
  PR Interval, Week 4: number analyzed (Participants) | 25 | 21 | 26
  PR Interval, Week 4 | -2.6 (7.32) | -3.1 (10.05) | 1.0 (15.22)
  PR Interval, Week 8: number analyzed (Participants) | 23 | 17 | 25
  PR Interval, Week 8 | -2.5 (10.40) | -3.1 (9.49) | 0.4 (15.88)
  QRS Duration, Week 4: number analyzed (Participants) | 25 | 21 | 27
  QRS Duration, Week 4 | -1.9 (5.17) | 2.1 (7.40) | 0.6 (8.38)
  QRS Duration, Week 8: number analyzed (Participants) | 23 | 17 | 25
  QRS Duration, Week 8 | -2.0 (4.99) | 1.0 (4.15) | 1.3 (8.35)

12. Secondary Outcome: Number of Participants With Shift From Baseline in Serum Laboratory Values (Clinical Chemistry)
Description: Serum laboratory parameters: Albumin, Alkaline phosphatase (AP), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Direct bilirubin, Total Bilirubin (T. Bilirubin), Calcium, Chloride, Carbon dioxide content/Bicarbonate (CO2/HCO3), Creatinine, Gamma glutamyl transferase (GGT), Glucose, Potassium, Sodium, Total protein (T. Protein), Urea/Blood urea nitrogen (BUN) and Uric acid were assessed. Baseline laboratory values were the latest values obtained on or before the participant's Baseline reference date. Unscheduled laboratory values were summarized as at-visit values only in the event that an at-visit laboratory value was missing. The values were presented as high, low or normal values shifted from Baseline value.
Time Frame: Baseline and up to follow up (post treatment 48 hours)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg
Number analyzed (Participants) | 27 | 22 | 28
Participants
  Albumin, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  Albumin, Week 4, high to normal | 2 | 1 | 1
  Albumin, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  Albumin, Week 4, normal to high | 1 | 2 | 0
  Albumin, Week 4, low to normal: number analyzed (Participants) | 25 | 21 | 26
  Albumin, Week 4, low to normal | 1 | 0 | 0
  Albumin, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  Albumin, Week 8, high to normal | 1 | 1 | 1
  Albumin, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  Albumin, Week 8, normal to high | 1 | 1 | 1
  Albumin, Week 8, low to normal: number analyzed (Participants) | 22 | 17 | 25
  Albumin, Week 8, low to normal | 1 | 0 | 0
  AP, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  AP, Week 4, high to normal | 0 | 0 | 1
  AP, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  AP, Week 4, normal to high | 0 | 0 | 1
  AP, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  AP, Week 8, high to normal | 0 | 0 | 1
  ALT, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  ALT, Week 4, high to normal | 1 | 0 | 0
  ALT, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  ALT, Week 4, normal to high | 1 | 1 | 1
  ALT, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  ALT, Week 8, high to normal | 2 | 0 | 0
  ALT, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  ALT, Week 8, normal to high | 0 | 1 | 1
  AST, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  AST, Week 4, normal to high | 0 | 1 | 2
  AST, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  AST, Week 8, normal to high | 0 | 1 | 0
  T. Bilirubin, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  T. Bilirubin, Week 4, normal to high | 2 | 1 | 2
  T. Bilirubin, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  T. Bilirubin, Week 4, high to normal | 0 | 0 | 4
  T. Bilirubin, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  T. Bilirubin, Week 8, high to normal | 2 | 0 | 4
  T. Bilirubin, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  T. Bilirubin, Week 8, normal to high | 0 | 1 | 2
  Calcium, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  Calcium, Week 4, high to normal | 1 | 0 | 0
  Calcium, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  Calcium, Week 4, normal to high | 1 | 0 | 1
  Calcium, Week 4, low to normal: number analyzed (Participants) | 25 | 21 | 26
  Calcium, Week 4, low to normal | 1 | 0 | 0
  Calcium, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  Calcium, Week 8, high to normal | 1 | 0 | 0
  Calcium, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  Calcium, Week 8, normal to high | 2 | 0 | 2
  Calcium, Week 8, low to normal: number analyzed (Participants) | 22 | 17 | 25
  Calcium, Week 8, low to normal | 1 | 0 | 0
  Chloride, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  Chloride, Week 4, high to normal | 1 | 0 | 0
  Chloride, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  Chloride, Week 4, normal to high | 1 | 2 | 0
  Chloride, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  Chloride, Week 8, high to normal | 1 | 0 | 0
  Chloride, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  Chloride, Week 8, normal to high | 1 | 0 | 0
  CO2/HCO3, Week 4, normal to low: number analyzed (Participants) | 25 | 21 | 26
  CO2/HCO3, Week 4, normal to low | 2 | 0 | 1
  CO2/HCO3, Week 4, low to normal: number analyzed (Participants) | 25 | 21 | 26
  CO2/HCO3, Week 4, low to normal | 2 | 3 | 2
  CO2/HCO3, Week 8, normal to low: number analyzed (Participants) | 22 | 17 | 25
  CO2/HCO3, Week 8, normal to low | 1 | 0 | 2
  CO2/HCO3, Week 8, low to normal: number analyzed (Participants) | 22 | 17 | 25
  CO2/HCO3, Week 8, low to normal | 2 | 3 | 1
  Creatinine, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  Creatinine, Week 4, normal to high | 1 | 0 | 0
  Creatinine, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  Creatinine, Week 8, normal to high | 1 | 0 | 0
  GGT, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  GGT, Week 4, high to normal | 0 | 0 | 1
  GGT, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  GGT, Week 4, normal to high | 0 | 0 | 1
  GGT, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  GGT, Week 8, high to normal | 0 | 0 | 1
  GGT, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  GGT, Week 8, normal to high | 0 | 0 | 2
  Glucose, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  Glucose, Week 4, high to normal | 1 | 2 | 1
  Glucose, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  Glucose, Week 4, normal to high | 3 | 2 | 2
  Glucose, Week 4, low to normal: number analyzed (Participants) | 25 | 21 | 26
  Glucose, Week 4, low to normal | 1 | 0 | 1
  Glucose, Week 4, normal to low: number analyzed (Participants) | 25 | 21 | 26
  Glucose, Week 4, normal to low | 0 | 1 | 0
  Glucose, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  Glucose, Week 8, high to normal | 2 | 1 | 3
  Glucose, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  Glucose, Week 8, normal to high | 2 | 4 | 1
  Glucose, Week 8, low to high: number analyzed (Participants) | 22 | 17 | 25
  Glucose, Week 8, low to high | 1 | 0 | 0
  Glucose, Week 8, low to normal: number analyzed (Participants) | 22 | 17 | 25
  Glucose, Week 8, low to normal | 0 | 0 | 1
  Potassium, Week 4, low to normal: number analyzed (Participants) | 25 | 21 | 26
  Potassium, Week 4, low to normal | 1 | 0 | 0
  Potassium, Week 8, low to normal: number analyzed (Participants) | 22 | 17 | 25
  Potassium, Week 8, low to normal | 1 | 0 | 0
  Sodium, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  Sodium, Week 4, high to normal | 0 | 1 | 1
  Sodium, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  Sodium, Week 4, normal to high | 0 | 1 | 0
  Sodium, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  Sodium, Week 8, high to normal | 0 | 1 | 1
  T. Protein, Week 8, low to normal: number analyzed (Participants) | 22 | 17 | 25
  T. Protein, Week 8, low to normal | 1 | 0 | 0
  Urea/BUN, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  Urea/BUN, Week 4, high to normal | 0 | 0 | 1
  Urea/BUN, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  Urea/BUN, Week 4, normal to high | 0 | 0 | 1
  Urea/BUN, Week 4, low to normal: number analyzed (Participants) | 25 | 21 | 26
  Urea/BUN, Week 4, low to normal | 0 | 0 | 1
  Urea/BUN, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  Urea/BUN, Week 8, high to normal | 0 | 0 | 1
  Uric acid, Week 4, high to normal: number analyzed (Participants) | 25 | 21 | 26
  Uric acid, Week 4, high to normal | 1 | 1 | 0
  Uric acid, Week 4, normal to high: number analyzed (Participants) | 25 | 21 | 26
  Uric acid, Week 4, normal to high | 1 | 0 | 2
  Uric acid, Week 4, low to normal: number analyzed (Participants) | 25 | 21 | 26
  Uric acid, Week 4, low to normal | 1 | 0 | 0
  Uric acid, Week 4, normal to low: number analyzed (Participants) | 25 | 21 | 26
  Uric acid, Week 4, normal to low | 0 | 0 | 1
  Uric acid, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  Uric acid, Week 8, normal to high | 1 | 0 | 0
  Uric acid, Week 8, low to normal: number analyzed (Participants) | 22 | 17 | 25
  Uric acid, Week 8, low to normal | 1 | 0 | 0
  Uric acid, Week 8, high to normal: number analyzed (Participants) | 22 | 17 | 25
  Uric acid, Week 8, high to normal | 0 | 1 | 0
  Uric acid, Week 8, normal to low: number analyzed (Participants) | 22 | 17 | 25
  Uric acid, Week 8, normal to low | 0 | 0 | 1

13. Secondary Outcome: Number of Participants With Shift From Baseline in Additional Lab Parameters (Free T3, Prostate Specific Antigen [PSA], Thyroid Stimulating Hormone [TSH] and Total Testosterone)
Description: Baseline laboratory values were the latest values obtained on or before the participant's Baseline reference date. Unscheduled laboratory values were summarized as at-visit values only in the event that an at-visit laboratory value was missing. The values were presented as high, low or normal values shifted from Baseline value.
Time Frame: Baseline and up to follow up (post treatment 48 hours)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Groups:
- GSK557296 50mg: Participants received one 50 mg tablet of study drug and two placebo tablets approximately one hour prior to planned SI, once in a 24-hour time period, on-demand for 8 weeks
- GSK557296 150mg: Participants received three 50 mg tablets of study drug approximately one hour prior to planned SI, once in a 24-hour time period, on-demand for 8 weeks.
Arm/Group | Placebo | GSK557296 50mg | GSK557296 150mg
Number analyzed (Participants) | 25 | 22 | 28
Participants
  Free T3, Week 4, high to nomal: number analyzed (Participants) | 25 | 21 | 26
  Free T3, Week 4, high to nomal | 0 | 1 | 0
  Free T3, Week 8, high to nomal: number analyzed (Participants) | 22 | 17 | 25
  Free T3, Week 8, high to nomal | 0 | 1 | 0
  TSH, Week 4, normal to low: number analyzed (Participants) | 25 | 21 | 25
  TSH, Week 4, normal to low | 0 | 1 | 0
  TSH, Week 8, normal to high: number analyzed (Participants) | 22 | 17 | 25
  TSH, Week 8, normal to high | 0 | 1 | 0
  Testosterone, Week 8, normal to low: number analyzed (Participants) | 22 | 17 | 25
  Testosterone, Week 8, normal to low | 1 | 1 | 1

14. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment. On-treatment adverse events were those started on or after the first dose of study medication and on or before the last dose of study medication.
Time Frame: Baseline and up to follow up (post treatment 48 hours)
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg
Number analyzed (Participants) | 25 | 22 | 28
Participants
  Any AEs | 8 | 6 | 10
  Any SAEs | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Dose/Exposure Response Relationship Using PK/Pharmacodynamics (PD) Modeling
Description: The relationship between plasma concentrations of GSK557296 and selected endpoints were planned to be explored using appropriate PK/PD models.
Time Frame: Up to Week 8
Population: ITT Population. Data was not collected for this outcome measure.
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All SAEs and non SAEs were collected through out the study treatment (8 weeks) and up to follow up (post treatment 48 hours)
Description: On-treatment SAEs and AEs are reported for safety Population, which consisted of all participants randomized to study treatment who received at least one dose of study drug.
Arm/Group | Placebo | GSK557296 50 mg | GSK557296 150 mg
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22 | 0/28
Other Adverse Events (participants affected / at risk) | 8/25 | 6/22 | 10/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | GSK557296 50 mg (N=22) | GSK557296 150 mg (N=28)
Headache (Nervous system disorders) | 3 | 3 | 5
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 2 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 1 | 0
Irritability (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Genital discomfort (Reproductive system and breast disorders) | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.